CLINICAL TRIAL: NCT05840081
Title: Effect of Full-Fat and Fat-Free Dairy, With and Without Fermentation, on Fecal Microbiome, Fecal and Serum Metabolome, and Host Cardiometabolic Risk Status
Brief Title: Dairy Fat and Fermentation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Alice Lichtenstein, D.Sc., Tufts University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3070
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Diseases; Microbial Colonization; Inflammation
Keywords: gut microbiome; gut microbiota; yogurt; milk; heart disease
MeSH Terms: conditions — Heart Diseases; Communicable Diseases; Inflammation | interventions — Milk

STUDY DESIGN:
Intervention Model Description: randomized crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Full-fat milk beverage (Experimental): Beverage made with full-fat milk
  Interventions: Other: Milk or yogurt beverage
- Fat-free milk beverage (Experimental): Beverage made with fat-free milk
  Interventions: Other: Milk or yogurt beverage
- Full-fat yogurt beverage (Experimental): Beverage made with full-fat yogurt
  Interventions: Other: Milk or yogurt beverage
- Fat-free yogurt beverage (Experimental): Beverage made with fat-free yogurt
  Interventions: Other: Milk or yogurt beverage

INTERVENTIONS:
Other: Milk or yogurt beverage — Commercially available milk or yogurt (depending on experimental arm) will be incorporated into flavored drinks/smoothies to minimize perceived differences among these items, preserving the double-blind nature of the study design.

SUMMARY:
The purpose of the study is to compare the effect of consuming full-fat (regular) and fat-free (skim) milk, as well as full-fat and fat-free yogurt (a fermented dairy product), on microorganisms in your gut as well as the products produced by the gut microbes. We will also determine whether consuming these dairy products affects risk factors for heart disease.The findings of the study will help us determine if heart disease risk factors are modified by the fat content and fermentation of milk. The results may facilitate refinement of public health dietary guidance for cardiovascular disease risk reduction.

DETAILED DESCRIPTION:
A randomized-controlled cross-over trial will be conducted to compare the effect of two servings per day of full-fat and fat-free milk, and full-fat and fat-free yogurt (hence forth referred to as dairy food items) on the gut microbiome, fecal and serum metabolome, and determine their relation to cardiometabolic risk factors (CMRF) and functional pathways associated with the differences identified. Participants will be provided with 2 servings per day of the test dairy products and requested not to consume additional bovine (cow) milk or yogurt during each 3-week diet phase.They will be allowed to use dairy substitutes such as plant-based milk alternatives and consume other types of dairy products (e.g. cheese).

The study consists of four diet phases: fat-free milk phase, full-fat milk phase, fat-free yogurt phase and full-fat yogurt phase. Each diet phase is 3 weeks in duration, separated by a 2 week break. Participants will be provided with 2 servings of a dairy based food item per day specific to their assigned phase and asked to consume them at two separate times during the day - morning and evening. Weight, waist circumference and blood pressure will be measured, blood and stool samples will be collected, and participants will complete two 24-hr food recall questionnaires during each phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age >50 years
2. Men and postmenopausal women
3. BMI >25 and <35 kg/m2
4. No milk allergy, lactose intolerance or adherence to vegan or other dietary pattern that excludes dairy products
5. Non-smoker
6. Usual pattern of bowel movements at least every other day.

Exclusion Criteria:

1. Women and men <50 years
2. Women, pre- or peri-menopausal
3. BMI <25 and >35 kg/m2
4. Current smokers or former smoker who quit < 6 months
5. Use of nicotine replacement products within last 6 months
6. Replacement or gender affirming hormonal therapy use
7. Weight gain of >15 pounds within last 6 months
8. Infrequent bowel movements
9. History of anemia within past 2 years or confirmation of anemia at first study visit
10. Blood donation within last 2 months
11. Untreated hypertension
12. Oral antibiotics use within 2 weeks of study entry
13. Steroid use (including dental prophylaxis use within 2 wks prior to or during study, except non-prescription topical and nasal steroids, e. g. Flonase)
14. Use of lipid lowering medications
15. Chronic use of aspirin, non-steroidal anti-inflammatory medications (NSAIDS), laxatives, anti-diarrheal medication
16. Regular use (>2 times per week) of acid lowering medication: antacids, proton pump inhibitors, or H2 Blockers.
17. Use of dietary supplements other than multi-vitamins, including pre- and probiotics, within 2 months of study entry
18. Milk allergy, lactose intolerance or adherence to vegan or other dietary patterns that exclude dairy products
19. Colonoscopy within 3 weeks of study entry or during study period
20. Diagnosis of malabsorption, inflammatory bowel disease (ulcerative colitis or Crohn's Disease), cirrhosis, history of gastrointestinal resection (other than appendectomy), chronic pancreatitis or any other chronic GI disease that in the opinion of the study physician would alter the study results
21. Chronic heart, liver, thyroid, renal or kidney disease
22. Type I or type II diabetes
23. Alcohol consumption >7 drinks/week for women and >14 drinks/week for men
24. Inadequate refrigerator storage capacity to store 21 8-oz containers of milk or yogurt
25. Participation in other dietary intervention research study during the same time
26. No social security number
27. Not willing to commit to adhering to the protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
gut microbiome | 3 weeks
  Determine the effects of dairy fat in milk, with and without fermentation, on gut microbiome
fecal metabolome | 3 weeks
  Determine the effects of dairy fat in milk, with and without fermentation, on fecal metabolome
serum metabolome | 3 weeks
  Determine the effects of dairy fat in milk, with and without fermentation, on serum metabolome

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D. Sc., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging, Boston, Massachusetts, United States